CLINICAL TRIAL: NCT01344551
Title: Effects of Cocoa Flavanols on Human Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor of Nutritional Medicine, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: UReading-2011-02
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Neural Degeneration
MeSH Terms: conditions — Nerve Degeneration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Flavanol (Active Comparator): High Flavanol cocoa drink containing 495mg cocoa
  Interventions: Dietary Supplement: Cocoa Drink
- Low Flavanol (Placebo Comparator): Low Flavanol cocoa drink (23mg)
  Interventions: Dietary Supplement: Cocoa Drink

INTERVENTIONS:
Dietary Supplement: Cocoa Drink — High Flavanol (495mg) Low Flavanol (23mg) Matched for macro and micro nutrients

SUMMARY:
To determine the acute and chronic effects of cocoa derived flavonoids on cognitive function in healthy older adults.

DETAILED DESCRIPTION:
This is a randomised controlled double blind cross over study investigating the acute effects of high flavanol (495mg) compared to low flavanol (23mg)cocoa drink on cognitive function in a healthy older adult population (n=60). The primary outcome measure of this study is to determine the effects of the flavanol intervention on cognitive measures of executive function and attention and the secondary measures of blood pressure and to determine whether any observed effects are paralleled by plasma flavanol levels.

ELIGIBILITY:
Inclusion Criteria:

* Aged 62 - 75 years
* A signed consent form

Exclusion Criteria:

* Blood pressure > 160/90 mmHg
* Haemoglobin (anaemia marker) < 125 g/l
* Gamma GT (liver enzymes) > 80 IU/l
* Had suffered a myocardial infarction or stroke in the previous 12 months
* Suffers from any gastrointestinal/stomach disorder
* Suffers from any blood-clotting disorder
* On medication for hypertension
* Suffers from any metabolic disorders (e.g. diabetes or any other endocrine or liver diseases)
* Depression or major mental illness
* Any dietary restrictions or on a weight reducing diet
* Drinking more than 21 units per week
* On any medication affecting blood clotting
* Smoking
* Vegans

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Executive function - attention | change from baseline to 2 hours

SECONDARY OUTCOMES:
Blood pressure | change from baseline to 2 hours
Plasma flavanols | change from baseline to 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Spencer, PhD, Principal Investigator — University of Reading; Laurie Butler, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom